CLINICAL TRIAL: NCT04906967
Title: A Comparative Study of Modified Sural Flap and Anterolateral Thigh Flap in Soft Tissue Reconstruction of Lower Extremity
Brief Title: Sural Flap and Anterolateral Thigh Flap in Tissue Reconstruction Around the Ankle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Faisal Esmael Mahmoud, Assistant lecturer in orthopedic department,faculty of medicine,sohag university,Sohag Governorate, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tissue coverage around ankle
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified sural flap (Active Comparator): modified sural flap used to cover soft tissue defect around ankle
  Interventions: Procedure: flaps
- anterolateral thigh flap (Active Comparator): anterolateral thigh flap used to cover soft tissue defect around ankle
  Interventions: Procedure: flaps

INTERVENTIONS:
Procedure: flaps — coverage of soft tissue defect around ankle

SUMMARY:
The aim of the study is to evaluate the outcomes of coverage of soft tissue defects of leg and foot by modified sural flap versus anterolateral thigh flap

DETAILED DESCRIPTION:
The leg and foot contain a thin subcutaneous layer and few muscles, thus the tibia and tendons can easily become exposed due to trauma. Therefore leg and foot injuries are often associated with a loss of soft tissues and exposed fractures.

one of the following reconstructive options are chosen:

1. The defect is allowed to heal by secondary intention.
2. The wound is closed primarily.
3. A split or full thickness skin graft and or neodermis is applied.
4. A local random flap or propeller flap is transposed or advanced.
5. A pedicled or island flap is transferred.
6. A microvascular free flap is transferred. The method of soft tissue reconstruction chosen hinges on the patient's medical condition, the surgeon's experience, the size of the wound, the vascular status of the foot and the exposed structures the skin in this region has low flexibility and the subcutaneous circulation does not allow the use of long randomized flaps, the task of finding flaps to cover bones or tendons in wounds with cutaneous loss in the legs and feet is difficult.

The sural flap acts as an axial flap and has 3 sources of nutrition,the vascular plexus of the deep fascia, the medial superficial sural artery which follows the medial sural nerve and the arteries that follow the minor saphenous vein. Venous return is ensured by the minor saphenous vein which may be used as a distal pedicle to provide reverse flow.

sural flap has the advantages of easy and quick harvesting without sacrificing major arteries and can be done in one stage operation.

In the other hand,Since introduction of the anterolateral thigh flap in 1984 by Song et al it has gained widespread popularity, especially in Asian countries, where it has replaced the radial forearm flap as being the workhorse in head and neck surgery.

Anterolateral thigh flaps have been introduced also in lower extremity reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* • patients aging 5 to 70 years.

  * Defect at the lower leg ,ankle or foot
  * Palpable distal pulse

Exclusion Criteria:

* • Peripheral vascular disease

  * Underling bone osteomyelitis
  * Unhealthy skin of posterior or lateral aspect of leg.
  * Vascular injury.
  * Patients with chronic diseases
  * Patients associated with vital organ injuries
  * Patients unfit to surgery

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Viability of the flap | baseline
  Viability of flap detected by numbers of flap survived in each group
Size of defect covered(size of the flap) | Baseline
  Detected by measuring the length and width in cms
Resistance to infection | Baseline
  Detected by numbers of flabs in each group that resist infection

REFERENCES:
- [Background] Noaman HH, Soroor YO. Foot salvage using microsurgical free muscle flaps in severely crushed foot with soft tissue defects. Injury. 2019 Dec;50 Suppl 5:S17-S20. doi: 10.1016/j.injury.2019.10.040. Epub 2019 Oct 23. PMID 31785835
- [Background] Battiston B, Antonini A, Tos P, Daghino W, Massazza G, Riccio M. Microvascular reconstructions of traumatic-combined tissue loss at foot and ankle level. Microsurgery. 2011 Mar;31(3):212-7. doi: 10.1002/micr.20863. Epub 2011 Feb 23. PMID 21351140